CLINICAL TRIAL: NCT00497068
Title: Tobacco Use in Opioid Agonist Treated Pregnant Women
Acronym: ROSE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Hendree E. Jones, Adjunct Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA012403 (NIH); R01DA012403 (NIH); DPMCDA
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Nicotine Dependence
Keywords: smoking; pregnancy; neonatal abstinence syndrome
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Neonatal Abstinence Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- tobacco abstinent contingent voucher (Experimental): Tobacco abstinent contingent voucher condition
  Interventions: Behavioral: tobacco abstinent contingent
- non-contingent (Experimental): Participants receive vouchers non-contingent upon tobacco use status
  Interventions: Behavioral: non-contingent
- no voucher (Other): This is the standard care intervention
  Interventions: Behavioral: control

INTERVENTIONS:
Behavioral: tobacco abstinent contingent — Participants receive vouchers wiht monetary rewards for providing breath samples that show tobacco smoking abstinence
  Arms: tobacco abstinent contingent voucher
Behavioral: non-contingent — Participants receive vouchers regardless of tobacco use status
  Arms: non-contingent
Behavioral: control — this group receives no vouchers
  Arms: no voucher

SUMMARY:
The primary objective of the proposed study is to evaluate the efficacy of tobacco abstinence-contingent voucher incentives versus non-tobacco abstinence-contingent incentives for reducing or eliminating tobacco use during pregnancy in methadone treated women. In addition, the impact that this intervention has in reducing the incidence and severity of methadone associated neonatal abstinence syndrome will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pregnancy
* Treatment entry at or before 31 weeks EGA
* Expected to enter drug-free outpatient modality at CAP
* Placed on methadone pharmacotherapy
* Nicotine dependent
* Sufficient literacy and understanding for assessment procedures
* Expected availability for study duration (e.g., complete inpatient stay)
* Able and willing to provide informed consent
* At least 18 years of age
* Confirmed smoker of 10 or more cigarettes

Exclusion Criteria:

* Not pregnant
* EGA of 32 weeks or greater
* 17 years of age or younger
* Undergoing detoxification (non-methadone treatment)
* Unable to provide informed consent
* Currently receiving nicotine replacement products (NRT)
* Current diagnosis of alcohol or benzodiazepine dependence
* Severe medical or psychiatric concomitant conditions that would interfere with treatment or require extended hospitalization.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2005-01; Primary Completion 2009-09 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Percent of tobacco-free urine samples submitted and Neonatal Abstinence Score | from treatment entry until 6 weeks post-partum

SECONDARY OUTCOMES:
tobacco use measures • treatment compliance• Neonatal measures include:Birth parameters | from treatment entry to 6 weeks posrt-partum

CONTACTS AND LOCATIONS:
Overall Officials: Hendree E Jones, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Center for Addiction and Pregnancy, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Tuten M, Svikis DS, Keyser-Marcus L, O'Grady KE, Jones HE. Lessons learned from a randomized trial of fixed and escalating contingency management schedules in opioid-dependent pregnant women. Am J Drug Alcohol Abuse. 2012 Jul;38(4):286-92. doi: 10.3109/00952990.2011.643977. Epub 2012 Feb 22. PMID 22352784